CLINICAL TRIAL: NCT03963700
Title: Genomic Profile and Tumor Immune Attack in Paraneoplastic Neurological Syndromes (PNS)
Brief Title: Tumor Characteristics in Patients With Paraneoplastic Neurological Syndromes (PNS)
Acronym: GenePNS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: GenePNS
Record Dates: First submitted 2019-04-26; First posted 2019-05-28 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Paraneoplastic Syndromes; Neurologic Disorder; Immune System and Related Disorders; Tumor Genetics
MeSH Terms: conditions — Neoplasms; Paraneoplastic Syndromes; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with Paraneoplastic neurological syndromes: Cancer patients with Paraneoplastic neurological syndromes presenting various autoimmune anomalies:
  * Anti-Hu also known as anti-Neuron specific cell Nuclear Antibodies (anti-ANNA1) (350 patients), uncommon form of brain inflammation associated with an underlying cancer
  * anti-Yo (130 patients), antibody associated with paraneoplastic cerebellar degeneration
  * anti-Ma2 (50 patients), antibody associated with paraneoplastic encephalitis
  * anti-N-methyl-d-aspartate (NMDA) Receptor (350 patients), autoimmune disorder in which antibodies attack N-methyl-D-aspartate-type glutamate receptors
  * anti-gamma-aminobutyric acid-B (GABAb) receptor (35 patients), autoimmune disorder in which antibodies attack gamma-aminobutyric acid-B receptors
  * anti-alpha-amino-3-hydroxy-5-methylisoxazole-4-propionic acid (AMPA) receptor (15 patients), autoimmune disorder in which antibodies attack alpha-amino-3-hydroxy-5-methylisoxazole-4-propionic acid receptors
  * without antibodies (50 patients).

SUMMARY:
Paraneoplastic neurological syndromes (PNS) are immune-mediated complications of cancer that can affect any part of the central or peripheral nervous system.

PNS occurs at the intersection between immune system and the tumor, where a combination of genetical and environmental factors may play a role.

Mechanisms leading to immune tolerance breakdown and autoimmunity in PNS remain largely unknown, and this reflects in an unsatisfactory repertoire of treatments available. Moreover, a better understanding of the biological mechanisms underlying PNS would allow a more precise identification of the modalities that permit PNS patients to have a better oncological prognosis than cancer patient without PNS, with obvious repercussions in clinical oncology.

To this effect, an extremely innovative approach involves directly exploring the tumoral tissue of patients suffering from specific PNS via genomic and transcriptomic analysis.

The study team hypothesizes that antigen ectopic expression by tumour cells may contribute to the generation of PNS.

In the present study, the investigators will analyze the salient features of tumors associated with PNS, namely the histological and immune cells infiltrate characteristics, their transcriptomic profile, and mutational status of involved antigens.

ELIGIBILITY:
Inclusion Criteria:

* presence of well characterized antibodies in serum or cerebrospinal fluid;
* histologically proven cancer with available tumour sample;
* Paraneoplastic neurological syndrome (PNS) diagnosis according to the international guidelines;
* Age: at least 18 years old.

Exclusion Criteria:

* Absence of complete clinicopathological data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer and suspected Paraneoplastic neurological syndrome (PNS) whose sample was sent for analysis at the Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France, for paraneoplastic antibody study and then stored at the biobank Neurobiotec.
Sampling Method: Non-Probability Sample
Enrollment: 980 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of mutations in cancer genes coding for onconeural proteins and inflammatory response mediators. | 36 months
  Genetic alterations in tumors associated with Paraneoplastic neurological syndromes (PNS)

SECONDARY OUTCOMES:
Proportion of different immune cells in the tumor's immune infiltrate | 36 months
  Histological immune infiltrate characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jerome HONNORAT, PhD, Principal Investigator — Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France